CLINICAL TRIAL: NCT00445900
Title: Phase II Study of the Combination of Low-Dose Thalidomide, Prednisone, and Oral Cyclophosphamide ("TPC") in the Therapy of Myelofibrosis With Myeloid Metaplasia (MMM)
Brief Title: Thalidomide, Prednisone, and Cyclophosphamide in Treating Patients With Myelofibrosis and Myeloid Metaplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Ruben A. Mesa, M.D., Mayo Clinic
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000530973; P30CA015083 (NIH); MC028A (Other: Mayo Clinic Cancer Center); 1360-03 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2007-03-07; First posted 2007-03-09 (Estimated); Last update posted 2011-03-17 (Estimated); Status verified 2011-03

CONDITIONS: Chronic Myeloproliferative Disorders; Secondary Myelofibrosis
Keywords: primary myelofibrosis; essential thrombocythemia; polycythemia vera; secondary myelofibrosis
MeSH Terms: conditions — Myeloproliferative Disorders; Primary Myelofibrosis; Thrombocythemia, Essential; Polycythemia Vera | interventions — Cyclophosphamide; Prednisone; Thalidomide; Immunohistochemistry; Biopsy

INTERVENTIONS:
Drug: cyclophosphamide
Drug: prednisone
Drug: thalidomide
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Procedure: biopsy

SUMMARY:
RATIONALE: Giving thalidomide together with prednisone and cyclophosphamide may lessen symptoms caused by myelofibrosis and myeloid metaplasia.

PURPOSE: This phase II trial is studying the side effects and how well giving thalidomide together with prednisone and cyclophosphamide works in treating patients with myelofibrosis and myeloid metaplasia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the benefit of thalidomide, prednisone, and cyclophosphamide in alleviating disease-associated anemia, thrombocytopenia, and/or splenomegaly in patients with myelofibrosis with myeloid metaplasia (MMM).
* Determine the benefit of this regimen in palliating four hypercatabolic constitutional symptoms (i.e., weight loss, fatigue, drenching night sweats, and unexplained fevers) in these patients.
* Determine the toxicity profile of this regimen in these patients.

Secondary

* Determine the effect of this regimen on leukocyte count.
* Determine the effect of this regimen on bone marrow histology, including microvessel density and reticulin fibrosis.
* Determine the effect of this regimen on intramedullary and urinary markers of angiogenesis.
* Determine the effect of this regimen on circulating myeloid progenitor cells by quantifying CD34+ cells.

OUTLINE: Patients receive oral thalidomide, oral prednisone, and oral cyclophosphamide (TPC) once daily on days 1-28. Treatment repeats every 28 days for 3 courses. After 3 courses (3 months) of treatment, patients who respond to TPC therapy may receive oral thalidomide alone once daily for up to 3 months in the absence of disease progression or unacceptable toxicity.

Patients undergo bone marrow aspirate and biopsy prior to study entry, 6 months after starting therapy, and then every 6 months for up to 3 years. Samples are analyzed by microvessel density/angiogenesis studies (i.e., CD34 immunohistochemical and vascular endothelium-specific staining) to determine the effect of therapy on markers of bone marrow angiogenesis.

After completion of study therapy, patients are followed every 6 months for up to 3 years.

PROJECTED ACCRUAL: A total of 22 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed myelofibrosis with myeloid metaplasia (MMM) of any of the following subtypes:

  * Agnogenic myeloid metaplasia
  * Post-polycythemic myeloid metaplasia
  * Post-thrombocythemic myeloid metaplasia
* Must have 1 of the following MMM-related conditions:

  * Anemia, defined as hemoglobin < 10 g/dL

    * Iron deficiency must be excluded as cause
  * Thrombocytopenia, defined as platelet count < 100,000/mm³
  * Palpable hepatomegaly or splenomegaly
* No evidence of myelofibrosis-associated conditions in the bone marrow, including any of the following:

  * Metastatic carcinoma
  * Lymphoma
  * Myelodysplasia
  * Hairy cell leukemia
  * Mast cell disease
  * Acute leukemia (including M7 type)
  * Acute myelofibrosis
* No chromosomal translocation t(9:22) or bcr-abl as determined by bone marrow chromosome analysis or peripheral blood fluorescent in situ hybridization (FISH) analysis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-3
* Absolute neutrophil count ≥ 750/mm³
* Bilirubin ≤ 2 times upper limit of normal (ULN), unless elevation due to MMM
* AST ≤ 5 times ULN, unless elevation due to MMM
* Creatinine ≤ 2.5 mg/dL
* No uncontrolled infection, including tuberculosis

  * No known history of positive purified protein derivative (PPD) untreated by isoniazid therapy

    * Positive PPD with normal chest X-ray and completion of full-course isoniazid therapy allowed
* No federal medical center inmates or other incarcerated patients
* No peripheral neuropathy ≥ grade 2
* No comorbid condition in which the use of study therapy is felt to be potentially harmful
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 forms of effective contraception

PRIOR CONCURRENT THERAPY:

* No chemotherapy (e.g., hydroxyurea, myelosuppressive therapy) within the past 14 days
* Prior splenectomy for MMM allowed
* No concurrent hematopoietic growth factors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2004-10; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Confirmed response, defined as a complete or partial response in ≥ 1 of 3 response categories (i.e., anemia, thrombocytopenia, or splenomegaly or hepatomegaly)

SECONDARY OUTCOMES:
Constitutional symptom status and bone marrow morphology
Overall survival
Progression-free survival
Time to progression
Duration of response
Toxicity as measured by NCI CTC v 2.0

CONTACTS AND LOCATIONS:
Overall Officials: Ruben A. Mesa, MD, Study Chair — Mayo Clinic